CLINICAL TRIAL: NCT04428242
Title: Evaluation of the Retinal Health Monitoring System - Retinal Thickness Module in Subjects With Normal Macular Thickness and Subjects With Center-involving Macular Edema
Brief Title: Study Evaluating Retinal Health Monitoring System Thickness Module
Status: Withdrawn | Type: Observational
Why Stopped: COVD-19
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCT-202
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Macular Edema; Macular Degeneration
Keywords: Macular Edema, Wet AMD; Retinal Thickness; Diabetic Retinopathy, Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Group 1: Subjects with normal macular thickness in one or both eyes.
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT
- Group 2: Subjects with center-involving macular edema due to w/AMD in one or both eyes.
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT
- Group 3: Subjects with center-involving macular edema due to DR or RVO in one or both eyes.
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT

INTERVENTIONS:
Device: RHMS-RTM — Assessment of retinal thickness.
  Other Names: Handheld swept source (SS) optical coherence tomography (OCT)
Diagnostic Test: SD-OCT — Assessment of retinal structure.

SUMMARY:
Evaluate the ability and accuracy of the Retinal Health Monitoring System - Retinal Thickness Module (RHMS - RTM).

DETAILED DESCRIPTION:
Evaluation of the Retinal Health Monitoring System - Retinal Thickness Module in subjects with normal macular thickness and subjects with center-involving macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Corrected visual acuity (VA) of 20/100 or better, in the study eye(s)
2. Media clarity, undilated pupil size, OCT-B scans, axial length measurements in the study eye(s)
3. Able to perform self-testing of retinal thickness with the RHMS-RTM after training
4. Able and willing to give informed consent
5. Group 1:

   1. Macula with normal thickness [central subfield thickness (CST) below 305 microns as measured by SD-OCT] in at least one eye
   2. Patients with dry AMD are eligible for enrollment into Group 1
   3. No history of wet AMD, DR, or RVO in either eye
6. Group 2 and Group 3 (in at least one or the same eye):

   1. History of center-involving macular edema due to wet AMD (Group 2); or DR or RVO (Group 3)
   2. Macular edema on SD-OCT with CST ≥ 305 microns

Exclusion Criteria:

1. History of corneal refractive surgery, photorefractive keratectomy, radial keratotomy, in the study eye
2. History of epiretinal membrane, vitreomacular traction, or macular hole in the study eye(s)
3. Participation in any study using an investigational drug within 30 days or screening or investigational device within 60 days of screening
4. Refractive error: spherical equivalent of > 3 diopters of hyperopia or > 6 diopters of myopia, or > 2 diopters cylinder in the study eye(s)
5. History of photocoagulation laser scar or other retinal scar in the central 3 mm of the macula, in the study eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged ≥ 18 years old with normal macular thickness, center-involving macular edema due to wAMD, diabetic retinopathy or retinal vein occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the RHMS-RTM retinal thickness measurements | 1 day
  To evaluate the ability of the RHMS-RTM device to measure retinal thickness
RHMS-RTM repeatability | 1 day
  To assess repeatability of the RHMS-RTM device
Comparison of retinal thickness measurements between the RHMS-RTM and the SD-OCT | 1 month
  To evaluate the agreement of measurements by the RHMS-RTM and SD-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gregory, MD, Study Director — Kubota Vision Inc.
Locations (1):
- Retinal Consultants Medical Group, Inc, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided